CLINICAL TRIAL: NCT05695664
Title: Comparison of the Postoperative Analgesic Effects of Ibuprofen Versus Ketorolac in Patients Undergoing Orthopedic Surgery
Brief Title: Postoperative Analgesic Effects of Ibuprofen Versus Ketorolac in Patients Undergoing in Orthopedic Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Collaborators: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Fazal Hussain Shah, Consultant General Surgeon, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156/05/21
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Intravenous Drug Usage; Ibuprofen; Ketorolac; Knee Arthroscopy; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Ketorolac

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Experimental): patient received 800 mg of Ibuprofen IV
  Interventions: Drug: Ibuprofen 800 mg
- Ketorolac (Experimental): Patients received Keterolac 30 mg IV
  Interventions: Drug: Ketorolac Injection

INTERVENTIONS:
Drug: Ibuprofen 800 mg — Intravenous injection of ibuprofen 800 mg
  Arms: Ibuprofen
Drug: Ketorolac Injection — Intravenous injection of Ketorolac 30 mg
  Arms: Ketorolac

SUMMARY:
Objectives: To compare the postoperative analgesic effects of ibuprofen versus ketorolac in patients undergoing orthopedic surgery at Combined Military Hospital, Rawalpindi.

Study design: Randomized controlled trial Setting: Department of Anasthesiology, Combined military Hospital, Rawalpindi Duration of study:6 months (01st August 2021 to 31st January 2022) Material and methods: After ethical approval, 100 patients in randomly divided two equal groups (A and B) were selected. In group A, 800 mg IV ibuprofen while in group B, 30 mg IV ketorolac was given within 30 min of skin closure after orthopedic surgery. The pain was assessed via visual analogue scale postoperatively. The SPSS version 25 was used for analysis of data. P value ≤ 0.05 was considered as significant.

DETAILED DESCRIPTION:
INTRODUCTION Healthcare seeks to decrease postoperative pain to ensure better and faster postoperative mobilization.1 Postoperative pain pathways identify populations at risk for 30-day readmissions and emergency department visits that are not due to post discharge complications.2 Chronic pain is acknowledged as a disease per se, and addressing pain control expectations before discharge could reduce surgical readmissions.3 However, despite advances in perioperative protocols, pain remains a very frequent clinical symptom seen by orthopedic surgeons and a major reason for patients to seek medical assistance. Moreover, pain management after orthopedic procedures remains suboptimal for many patients.4 For instance, 37% of orthopedic patients reported their pain to be severe at its highest intensity, where postoperative pain remains a problem that requires consensus and joint efforts.5 Several modalities are available to alleviate the postoperative period, which range from nerve blocks to the use of various classes of drugs. Opioids have been widely used for pain relief. However, this class of drug is associated with a wide range of side effects, including a potential for developing drug dependence and addiction. On the other hand, non-steroidal anti-inflammatory drugs (NSAIDs), have been used widely for pain relief. NSAIDs are widely available as compared to opioids. NSAIDs also have several side effects, but a study has proven NSAIDs to be safe for controlling acute postoperative pain if they are used appropriately.6 Several studies have compared the different drugs belonging to the NSAID class in terms of their efficacy as postoperative analgesia. A study found no difference in pain and satisfaction between two groups of patients receiving either IV ketorolac or IV Ibuprofen as part of postoperative analgesia following urogynecological surgeries.7 However, patients who underwent laparotomies had less pain with Keterolac.8 In another study carried out on patients undergoing knee arthroscopies, preemptive use of Ibuprofen 800 mg was associated with less postoperative pain.9 Uribe et al. compared the postoperative analgesic effects of ibuprofen and ketorolac and discovered a difference in rescue analgesic use (55% vs. 83.9%), time to first rescue analgesic use (77.62 ± 33.03 vs. 55.78 ± 35.37 hours), and analgesic requirement in PACU (5.53 ± 5.89 vs. 19.92 ± 15.63 mg, p value 0.05).10 Postoperative pain is one of the principal concerns of surgeons and anesthesiologists, which leads to prolonged hospitalization and an increased analgesic requirement. Both factors expose the patient to hospital acquired infection and the untoward side effects of analgesics. As a result, a balanced or multimodal analgesia with adjuvant medications is required. It is important that, as anesthesiologists, we understand the effective method for pain suppression during orthopedic procedures. Therefore, this study is aimed at filling this knowledge gap. Data from this study would add information and serve as a baseline for the development of management guidelines for pain management.

METHODS AND MATERIALS After obtaining approval from the Ethical Committee / Institutional Review Board (IRB) (document no. 156/05/21), patients undergoing orthopedic surgeries were enrolled in the Department of Anesthesiology and Orthopedics at the Combined Military Hospital, Rawalpindi. The sample size for this randomized controlled trial (RCT) was 100 patients (50 patients in each group), which was calculated from a previous study by taking the frequencies of rescue analgesic use as (55% vs. 83.9%). 11 The power of the test was 90% with a 5% level of significance. The research lasted six months, from August 1, 2021, to January 31, 2022. All patients gave their informed written consent. The patients of either gender with an age range of 40-80 years and an ASA grade of 2 who were undergoing orthopedic surgeries for fractures of the radius, ulna, and wrist were included in the study. Patients with a history of adverse reactions to ibuprofen or ketorolac, a history of epilepsy, bronchial asthma, coronary artery disease, renal or hepatic impairments, or use of antiarrhythmic or analgesic medications in the last seven days were excluded. Age, gender, obesity (BMI > 27 kg/m2), history of smoking (10 or more cigarettes per day for at least 5 years or 5 or more cigarettes per day for at least 10 years), diabetes, and hypertension were registered before pre-operative evaluation of the patients to assess their fitness for anesthesia. The patients were labeled as diabetics when they were on anti-diabetic medication for at least 6 months or when there was lab evidence of HBA1c >6.5%, fasting blood sugar of >126 mg/dL, or a random blood sugar level of >200 mg/dL. Patients were classified as hypertensive if they had been taking anti-hypertensive medication for at least 6 months or if clinical evidence of blood pressure greater than 140/90 was found on at least two separate occasions at least two hours apart. All patients were randomly divided into two equal groups (A and B) by using the sealed envelope technique. All surgeries were done under standard general anesthesia. Patients were induced with propofol (2 mg/kg) and premedicated with fentanyl. Endotracheal intubation was facilitated by the muscle relaxant atracurium 0.5 mg/kg. Anesthesia was maintained with 50% O2, 50% air, 1 MAC isoflurane, and atracurium. The patients were mechanically ventilated to keep ETCO2 between 35 and 40 mmHg. In Group A, patients received an intravenous injection of 800 mg of Ibuprofen, while intravenous ketorolac (30 mg) was given to patients in Group B, approximately 30 minutes before the skin closure. All patients were extubated and transferred to the post-anesthesia care unit (PACU). The durations of the surgical procedure and anesthesia were documented. Another anesthesiologist on duty was deputed for follow-up with the patients. The patients were kept blind to the type of analgesic drug they received. The postoperative pain was measured by VAS at 3, 6, and 12 hours postoperatively. The VAS ranged from 0 to 10, with 0 representing no pain and 10 representing the maximum bearable pain. When the VAS score was > 4, the injection Tramadol 30 mg was given intravenously as a rescue analgesic. The frequency of patients requiring rescue analgesia, the time to start rescue analgesia, and the total dose of drug during the 12-hour postoperative period were noted in each group.

Statistical analysis: The data was analyzed by IBM, SPSS Version 20 registered for Microsoft Windows. The mean, standard deviation, and frequency/percentages were calculated for quantitative and qualitative data, respectively. Chi square and independent sample t-tests were used to compare postoperative analgesic parameters between both groups. The p value of <0.05 was taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender undergo orthopedic surgery were included in the study.
* ASA ≤ 2
* Age 40-80 years.
* Fracture Radius , Ulna, and wrist

Exclusion Criteria:

* Patients with history of adverse response from ketorolac and ibuprofen was not taken into the study.
* Patients with history of epilepsy.
* Patients with history of cardiac conduction defects.
* Patients on antiarrhythmic drugs or analgesics.
* Patients with H/O stroke, renal impairment, chronic obstructive pulmonary disease, asthma, chronic liver disease, hypothyroidism and CCF were excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 3, 6 and 12 hours in postoperative period
  Postoperative pain measured by visual analogue scale (VAS), in which 0 is no pain and 10 is the maximum possible bearable pain.
Rescue analgesia requirement | 12 hours in the postoperative period
  Inj. Ketorolac 30 mg as Rescue analgesic was used intravenouly when VAS was equal or more than 4

CONTACTS AND LOCATIONS:
Locations (1):
- Fazal Hussain, Bhakkar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greimel F, Maderbacher G, Zeman F, Grifka J, Meissner W, Benditz A. No Clinical Difference Comparing General, Regional, and Combination Anesthesia in Hip Arthroplasty: A Multicenter Cohort-Study Regarding Perioperative Pain Management and Patient Satisfaction. J Arthroplasty. 2017 Nov;32(11):3429-3433. doi: 10.1016/j.arth.2017.05.038. Epub 2017 May 26. PMID 28641966
- [Background] Hernandez-Boussard T, Graham LA, Desai K, Wahl TS, Aucoin E, Richman JS, Morris MS, Itani KM, Telford GL, Hawn MT. The Fifth Vital Sign: Postoperative Pain Predicts 30-day Readmissions and Subsequent Emergency Department Visits. Ann Surg. 2017 Sep;266(3):516-524. doi: 10.1097/SLA.0000000000002372. PMID 28657940
- [Background] Masala IF, Caso F, Sarzi-Puttini P, Salaffi F, Atzeni F. Acute and chronic pain in orthopaedic and rheumatologic diseases: mechanisms and characteristics. Clin Exp Rheumatol. 2017 May-Jun;35 Suppl 105(3):127-131. Epub 2017 Jun 29. PMID 28681710
- [Background] Lavie LG, Fox MP, Dasa V. Overview of Total Knee Arthroplasty and Modern Pain Control Strategies. Curr Pain Headache Rep. 2016 Nov;20(11):59. doi: 10.1007/s11916-016-0592-6. PMID 27655139
- [Background] Ramia E, Nasser SC, Salameh P, Saad AH. Patient Perception of Acute Pain Management: Data from Three Tertiary Care Hospitals. Pain Res Manag. 2017;2017:7459360. doi: 10.1155/2017/7459360. Epub 2017 Mar 28. PMID 28458592